CLINICAL TRIAL: NCT02734134
Title: One Stage Versus Two Stage For Periprosthetic Hip And Knee Infection
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: OrthoCarolina Research Institute, Inc. (Other)
Collaborators: The Cleveland Clinic (Other); Hospital for Special Surgery, New York (Other); Rothman Institute at Thomas Jefferson University (Unknown); Midwest Orthopaedics Rush University Medical Center (Unknown); Vanderbilt University (Other); Emory University (Other); University of Iowa (Other); Carilion Clinic (Other); University of Southern California (Other); Ochsner Health System (Other); Cleveland Clinic Florida (Other); University of Utah (Other); University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1106
Record Dates: First submitted 2016-03-23; First posted 2016-04-12 (Estimated); Last update posted 2025-04-28 (Actual); Status verified 2025-04

CONDITIONS: Surgical Site Infection
Keywords: Periprosthetic joint infection
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- One-stage exchange (Active Comparator): One surgery where the infected implants are removed and the hip or knee joint are 'washed out' before new joint replacement implants are re-implanted during the same surgical procedure.
  Interventions: Procedure: One-stage exchange joint replacement surgery
- Two-stage exchange (Active Comparator): Two surgeries; during the first surgery the infected implants are removed and a spacer is placed in the hip or knee joint in place of the implants. A second surgery to re-implant the hip or knee joint replacement implants is performed if and when the infection has cleared.
  Interventions: Procedure: Two-stage exchange joint replacement surgery

INTERVENTIONS:
Procedure: One-stage exchange joint replacement surgery
  Arms: One-stage exchange
Procedure: Two-stage exchange joint replacement surgery
  Arms: Two-stage exchange

SUMMARY:
The purpose of this study is to compare the outcomes of two different treatment options commonly used to manage periprosthetic joint infection (PJI), an infection around the artificial knee or hip.

DETAILED DESCRIPTION:
Total joint arthroplasty (TJA) is a very common and successful procedure, and is expected to become more prevalent in the upcoming years. However, despite its success, TJA is associated with some complications, including periprosthetic joint infection (PJI). PJI is a devastating complication that is associated with marked patient morbidity and mortality and is an immense economic burden. Although the rate of PJI following a TJA is low, the burden is rising exponentially due to health complications and treatment costs. There are two common types of surgical treatments that can be used to treat chronic PJI, a two-stage exchange arthroplasty and a one-stage exchange arthroplasty. During a two-stage exchange arthroplasty, the implants are removed, infected tissues are debrided and a temporary antibiotic impregnated spacer fashioned from polymethylmethacrylate is placed (stage one). Afterwards the patient undergoes many weeks of intravenous antibiotics, followed by reimplantation at a later date (stage two). During the time between the first and second stage of the revision patients are often immobile, experience severe pain due to a lack of functioning joint, and may experience systemic toxicity associated with the administration of antibiotics. In a one stage exchange arthroplasty, the infected prosthesis is removed, infected tissues are debrided, and a new prosthesis is reimplanted during the same procedure.

While the two-stage exchange arthroplasty is the preferred method of treatment for chronic PJI in North America, the one-stage exchange arthroplasty is the method of choice in Europe and some centers have reported comparable results in terms of success for one-stage exchange to two-stage exchange arthroplasty. However, there has been no randomized, prospective, controlled study to date that compares one-stage exchange to two-stage exchange arthroplasty. Because of the lack of comparative outcome reports, and the perceived higher rate of failure of one-stage exchange arthroplasty, surgeons in North America prefer to perform the traditional two-stage exchange arthroplasty for management of chronic PJI. Several teams have succeeded in performing a one-stage exchange arthroplasty in selected patients, but this procedure has not gained much popularity in the US.

The purpose of this study is to investigate the outcome of one-stage and two-stage exchange arthroplasty for the management of patients with chronic PJI. The hypothesis of this study is that one-stage exchange arthroplasty, if performed in the appropriate patient population, carries a similar success rate for the treatment of chronic PJI as two-stage exchange arthroplasty and avoids many of the problems associated with two-stage exchange arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years old
* Patients who speak English and are willing to sign the consent form
* Patients with chronic infection of a total knee or total hip arthroplasty, defined as:

  * A sinus communicating with the prosthesis
  * Two positive cultures obtained from the prosthesis
  * 3 of 5 criteria: (i) Elevated erythrocyte sedimentation rate (ESR) (>30mm/jr) and c-reactive protein (CRP) (>10mg/L) (ii) Elevated synovial leukocyte count (>3000 cells/µL) or change of ++ on leukocyte esterase strip (iii) Elevated synovial neutrophil percentage (>80%) (iv) One positive culture (v) Positive histological analysis of periprosthetic tissue (>5 neutrophils per high power field in 5 high power fields x400)
* Patients with a previous irrigation and debridement for periprosthetic infection

Exclusion Criteria:

* Culture negative infections whereby the infecting organism has not identified
* Patients with systemic sepsis who require emergent surgery
* Patients with extensive soft tissue involvement that would preclude the closure of the wound after reimplantation, if the patient were to undergo the one-stage exchange
* Patients with acute PJI or acute hematogenous PJI, defined as:

  * Presentation of systems <4 weeks from index procedure
  * Presentation of systems <4 week duration
* Fungal infections
* Resistant organisms not sensitive to available IV antibiotics, oral antibiotics, or heat stable antibiotic additives to bone cement with documented elution characteristics
* Revision surgery or previous two-stage reimplant
* HIV positive patients or patients on chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 343 (Actual)
Dates: Start 2016-05-18 (Actual); Primary Completion 2024-12 (Actual); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Recurrence of infection | 1 year following treatment
  The primary outcome measured will be the recurrence of infection by the same organism or reinfection with a new organism as determined by the criteria using the International Consensus Meeting on PJI (1 year follow-up).

SECONDARY OUTCOMES:
Health Related Quality of Health | 2 years following surgery
  All patients will complete the Veteran's Rand - 12 (VR-12) which is a general health measure. The VR-12 also yields a health utility measure that can be used to calculate quality-adjusted life years in an economic cost-utility analysis.
Patient-Reported Functional Outcomes | 2 years following surgery
  Hip patients will complete the Hip disability and Osteoarthritis Outcome Score (HOOS), Junior which is a region-specific measure of pain and function of the hip.
Patient-Reported Functional Outcomes | 2 years following surgery
  Knee patients will complete the Knee injury and Osteoarthritis Outcome Score (KOOS) Junior which is a region-specific measure of pain and function of the knee.

OTHER OUTCOMES:
Death | 2 years
  Death within two years of surgical treatment for periprosthetic joint infection.
Percentage of patients requiring surgical revision for causes other than infection | Two years
  Revision of prosthetic joint for causes other than infection (e.g. hematoma, spacer dislocation).

CONTACTS AND LOCATIONS:
Overall Officials: Thomas K Fehring, MD, Principal Investigator — Attending Hip & Knee Surgeon
Locations (5):
- United States (5):
  - Midwest Orthopaedics at Rush University Medical Center, Chicago, Illinois
  - Hospital for Special Surgery, New York, New York
  - OrthoCarolina Research Institue, Charlotte, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Rothman Institute at Thomas Jefferson University, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zmistowski B, Karam JA, Durinka JB, Casper DS, Parvizi J. Periprosthetic joint infection increases the risk of one-year mortality. J Bone Joint Surg Am. 2013 Dec 18;95(24):2177-84. doi: 10.2106/JBJS.L.00789. PMID 24352771
- [Background] Luu A, Syed F, Raman G, Bhalla A, Muldoon E, Hadley S, Smith E, Rao M. Two-stage arthroplasty for prosthetic joint infection: a systematic review of acute kidney injury, systemic toxicity and infection control. J Arthroplasty. 2013 Oct;28(9):1490-8.e1. doi: 10.1016/j.arth.2013.02.035. Epub 2013 Apr 8. PMID 23578491
- [Background] Nickinson RS, Board TN, Gambhir AK, Porter ML, Kay PR. The microbiology of the infected knee arthroplasty. Int Orthop. 2010 Apr;34(4):505-10. doi: 10.1007/s00264-009-0797-y. Epub 2009 May 21. PMID 19458950
- [Background] El Helou OC, Berbari EF, Marculescu CE, El Atrouni WI, Razonable RR, Steckelberg JM, Hanssen AD, Osmon DR. Outcome of enterococcal prosthetic joint infection: is combination systemic therapy superior to monotherapy? Clin Infect Dis. 2008 Oct 1;47(7):903-9. doi: 10.1086/591536. PMID 18754743
- [Background] Parvizi J, Zmistowski B, Adeli B. Periprosthetic joint infection: treatment options. Orthopedics. 2010 Sep 7;33(9):659. doi: 10.3928/01477447-20100722-42. PMID 20839679
- [Background] Parkinson RW, Kay PR, Rawal A. A case for one-stage revision in infected total knee arthroplasty? Knee. 2011 Jan;18(1):1-4. doi: 10.1016/j.knee.2010.04.008. Epub 2010 Aug 17. PMID 20719522
- [Background] von Foerster G, Kluber D, Kabler U. [Mid- to long-term results after treatment of 118 cases of periprosthetic infections after knee joint replacement using one-stage exchange surgery]. Orthopade. 1991 Jun;20(3):244-52. German. PMID 1876406
- [Background] Buechel FF, Femino FP, D'Alessio J. Primary exchange revision arthroplasty for infected total knee replacement: a long-term study. Am J Orthop (Belle Mead NJ). 2004 Apr;33(4):190-8; discussion 198. PMID 15132327
- [Background] Singer J, Merz A, Frommelt L, Fink B. High rate of infection control with one-stage revision of septic knee prostheses excluding MRSA and MRSE. Clin Orthop Relat Res. 2012 May;470(5):1461-71. doi: 10.1007/s11999-011-2174-6. Epub 2011 Nov 12. PMID 22081299
- [Background] Ure KJ, Amstutz HC, Nasser S, Schmalzried TP. Direct-exchange arthroplasty for the treatment of infection after total hip replacement. An average ten-year follow-up. J Bone Joint Surg Am. 1998 Jul;80(7):961-8. doi: 10.2106/00004623-199807000-00004. PMID 9698000
- [Background] Leunig M, Chosa E, Speck M, Ganz R. A cement spacer for two-stage revision of infected implants of the hip joint. Int Orthop. 1998;22(4):209-14. doi: 10.1007/s002640050244. PMID 9795805
- [Background] Pattyn C, De Geest T, Ackerman P, Audenaert E. Preformed gentamicin spacers in two-stage revision hip arthroplasty: functional results and complications. Int Orthop. 2011 Oct;35(10):1471-6. doi: 10.1007/s00264-010-1172-8. Epub 2010 Nov 30. PMID 21116817
- [Background] Berend KR, Lombardi AV Jr, Morris MJ, Bergeson AG, Adams JB, Sneller MA. Two-stage treatment of hip periprosthetic joint infection is associated with a high rate of infection control but high mortality. Clin Orthop Relat Res. 2013 Feb;471(2):510-8. doi: 10.1007/s11999-012-2595-x. PMID 22983683
- [Background] Diaz-Ledezma C, Higuera CA, Parvizi J. Success after treatment of periprosthetic joint infection: a Delphi-based international multidisciplinary consensus. Clin Orthop Relat Res. 2013 Jul;471(7):2374-82. doi: 10.1007/s11999-013-2866-1. Epub 2013 Feb 26. PMID 23440616
- [Background] Berry DJ, Harmsen WS, Cabanela ME, Morrey BF. Twenty-five-year survivorship of two thousand consecutive primary Charnley total hip replacements: factors affecting survivorship of acetabular and femoral components. J Bone Joint Surg Am. 2002 Feb;84(2):171-7. doi: 10.2106/00004623-200202000-00002. PMID 11861721
- [Background] Daigle ME, Weinstein AM, Katz JN, Losina E. The cost-effectiveness of total joint arthroplasty: a systematic review of published literature. Best Pract Res Clin Rheumatol. 2012 Oct;26(5):649-58. doi: 10.1016/j.berh.2012.07.013. PMID 23218429
- [Background] Aggarwal VK, Rasouli MR, Parvizi J. Periprosthetic joint infection: Current concept. Indian J Orthop. 2013 Jan;47(1):10-7. doi: 10.4103/0019-5413.106884. PMID 23531512